CLINICAL TRIAL: NCT05615896
Title: Data Collection With the P200TE and P200TxE in Diseased Eyes for Clinical Developments
Brief Title: Data Collection With the P200TE and P200TxE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is no longer required.
Sponsor: Optos, PLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OPT1037
Record Dates: First submitted 2021-06-21; First posted 2022-11-14 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Intervention Model Description: A
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- P200TxE Device First (Experimental)
  Interventions: Device: Imaging Session
- P200TE Device First (Experimental)
  Interventions: Device: Imaging Session

INTERVENTIONS:
Device: Imaging Session — Various scans will be captured on both devices

SUMMARY:
The primary objective is to collect OCT scans on a modified P200TxE and P200TE.

ELIGIBILITY:
Inclusion Criteria :

* Male or female volunteers 22 years of age or older who have full legal capacity to volunteer on the date the informed consent is signed;
* Volunteers who can follow the instructions by the clinical staff at the clinical site;
* Volunteers who agree to participate;
* Volunteers who have been diagnosed with retina pathology with intra-retinal and/or subretinal fluid present in the posterior pole region.

Exclusion Criteria:

* Volunteers unable to tolerate ophthalmic imaging;
* Volunteers with ocular media not sufficiently clear to obtain acceptable OCT images.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Collection of images | 1 year
  The primary endpoint will be the collection of OCT scans on the P200TE and P200TxE devices. The scans will be used by R&D for development of a de-noising algorithm as well as other possible developments.

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Consultants of Texas Research Centers, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No